## <u>Can You Reduce Diabetes Symptomatology by Becoming Your 'Best Possible Self'?: The Role of Stress and Resilience</u>

Informed Consent Form

Last Edited: 14/09/2018



Researcher: Ben Gibson (B.Gibson@2016.ljmu.ac.uk)

## LIVERPOOL JOHN MOORES UNIVERSITY CONSENT FORM

Can You Reduce Diabetes Symptomatology by Becoming Your 'Best Possible Self'?: The Role of Stress and Resilience

School of Natural Sciences and Psychology, Tom Reilly Building, Room 313, Byrom Street, Liverpool, L3 3AF.

| Dire | ector of Studies: Dr Kanayo Umeh ( <u>F.K.Ume</u> | h@ljmu.ac.uk) | | |
|---|---|---|---|---|
| 1. | I confirm that I have read and understood the information provided. I have had the opportunity to consider the information, ask questions, and have had these answered satisfactorily. | | | _ |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving a reason and that this will not affect my legal rights. | | | _ |
| 3. | I understand that any personal information collected during the study will be anonymised and will remain confidential. | | | _ |
| 4. | I agree to take part in this study. | | | _ |
| Nar | ne of Participant | Date | Signature | |
| Nar | ne of Researcher | Date | Signature | |